CLINICAL TRIAL: NCT05067413
Title: A Prospective Non-randomized Controlled Multi-center Study of Laparoscopic Intracorporeal Distal Rectal Transection by Using the Traditional Approach vs. Using Transanterior Obturator Nerve Gateway Approach for Ultralow Rectal Cancers
Brief Title: A Study on the Efficacy of a Novel Approach to Achieving Laparoscopic Distal Rectal Transection for Rectal Cancers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Peking University First Hospital (Other)
Collaborators: Shengli Oilfield Hospital (Other); The Second Affiliated Hospital of Baotou Medical College (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020149; 320.6750.2021-04-2 (Other Grant/Funding Number: Wu Jieping's Foundation Special for Clinical Research)
Record Dates: First submitted 2021-08-25; First posted 2021-10-05 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-09

CONDITIONS: Rectal Neoplasms Malignant
Keywords: Laparoscopic; Ultralow rectal cancer; Intersphincteric resection; Total mesorectal excision; Transanterior obturator nerve gateway; Distal rectal transection

STUDY DESIGN:
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Total mesorectal excision approach (Sham Comparator): Patients of the control group who are to receive the traditional approach-- total mesorectal excision approach to transect the distal rectum are assigned into this arm.
  Interventions: Procedure: Total mesorectal excision approach
- Transanterior obturator nerve gateway approach (Experimental): Patients of the experimental group who are to receive the novel approach-- transanterior obturator nerve gateway approach to transect the distal rectum are assigned into this arm.
  Interventions: Procedure: Transanterior obturator nerve gateway approach

INTERVENTIONS:
Procedure: Transanterior obturator nerve gateway approach — Distal rectal transection of cases in the experimental group will be performed using transanterior obturator nerve gateway approach
  Arms: Transanterior obturator nerve gateway approach
Procedure: Total mesorectal excision approach — Distal rectal transection of cases in the control group will be performed using total mesorectal excision approach
  Arms: Total mesorectal excision approach

SUMMARY:
The wide application of ISR and DST has greatly improved the anal preservation rate for low rectal cancers, but the technical difficulty has also been obviously increased because of the limited pelvic space. Although many scholars have tried to solve this problem, all the methods have failed to fundamentally solve the problem of "the oblique dissection" of the distal rectum. To solve the problem above, the director of this clinical trial has explored a new distal rectal resection method-- transanterior obturator nerve gateway approach. The purpose of this clinical trial is to prospectively collect and compare data on the patients' perioperative variables and postoperative functional and oncological outcomes of this novel approach with the traditional approach to confirm the safety and feasibility of this novel approach and its advantages over the traditional approach.

DETAILED DESCRIPTION:
Objective To confirm the safety, feasibility and advantages by comparing the perioperative variables, postoperative functional and oncological outcomes of patients with ultralow rectal cancer treated by laparoscopic traditional distal rectal dissection vs. by transanterior obturator nerve gateway approach.

Patients Patients with ultralow (≤5cm from the anal verge) rectal cancer who are to undergo laparoscopic radical resection (ISR- DST) without any contraindications of general anesthesia, surgery or chemotherapy. (See details in Eligibility part) Sample size Two groups are designed, patients who are to receive the traditional approach to transect the distal rectum are assigned to the control group, patients who are to receive the transanterior obturator nerve gateway approach to transect the distal rectum are assigned to the experimental group. 100 cases are to be enrolled for the experimental group and not less than 100 cases are to be enrolled for the controlled group.

Treatment If the participant match with the requirements for this study and agree to take part in it, once hospitalized, the participant will complete the established preoperative tests including blood routine, the comprehensive metabolic panel, blood coagulation function, tumor markers, blood type, infectious disease screening tests, chest, abdominal and pelvic CT (Computed Tomography) scan and MRI (Magnetic Resonance Imaging), colonoscopy, echocardiogram, pulmonary function, venous duplex ultrasound of legs. All male patients will be routinely asked to fill in the IIEF-5 (International Index of Erectile Function-5) sexual function scoring questionnaire preoperatively.

The following comprehensive treatment will be depended on the examination results:

Neoadjuvant therapy The treatment plan will be made in accordance with the NCCN (National Comprehensive Cancer Network) Guidelines for Diagnosis and Treatment of Colorectal Cancer (Version 1.2021).

Neoadjuvant chemoradiotherapy: Pelvis radiotherapy with a total dose of 50 Gy with 25 courses in 5 weeks. Neoadjuvant chemotherapy include single drug therapy: capecitabine (CAP, 1250 mg/m2, BID) or double drug therapy: oxaliplatin combined with capecitabine (CapeOX, oxaliplatin 130 mg/m2, day 1, capecitabine 1000mg/ m2, day 1 ~ 14, then rest for 7 days, repeated every 3 weeks) or three-drug therapy (mFOLFOX6, oxaliplatin 85 mg/ m2 intravenous infusion for 2 hours, leucovorin calcium 400 mg/m2 intravenous infusion for 2 hours, 5-FU (fluorouracil) 400 mg/m2 intravenous infusion for 1 day, Then 1200 mg/ m2/d×2 days of continuous intravenous infusion with a total of 2400mg/m2 for 46 ~ 48 hours, repeated every 2 weeks.

Abdominal and pelvic MRI and contrast enhanced CT will be routinely performed 6 to 8 weeks after neoadjuvant therapy to confirm the extent of tumor regression without new-found distant metastasis. Those whose clinical stage after neoadjuvant therapy changes from T4 to T3 will be seen as eligible in this study.

Surgical treatment Preoperative preparation

1) Patients older than 60 years old or having a smoking history for over 10 years will receive lung ventilation training and atomization treatment for 3 days. 2) Intestinal preparation will be done with oral cathartic medications 12-24 hours before surgery. 3) Prophylactic antibiotics will be given once anesthesia is begun, the second antibiotics will be given if the operation lasts for over 3 hours. 4）Urethral catheterization will be routinely done preoperatively. 5）If the patient refuses to accept the novel approach before surgery, they will be directly enrolled in the traditional group. If both approaches are acceptable to the patient, the decision whether to use the novel approach will be made according to the intraoperative conditions (see operating procedures below).

Operating procedures General anesthesia; Modified lithotomy position; Establishment of pneumoperitoneum: Place a trocar 1cm above the umbilicus through which to establish pneumoperitoneum and keep the abdominal pressure as 12mmHg (millimeters of mercury).

Trocar placement: above the umbilicus (trocar C, 10 mm), upper right and left quadrants (trocars B and D, 5 mm), lower right quadrant (trocar A, 12 mm), lower left quadrant (trocar E, 5 mm), the midpoint between the pubic symphysis and umbilicus (trocar F, 5 mm).

Abdominal exploration: Explore the abdominal cavity in accordance with the principle of non-contact, from far to near step by step, explore the tumor finally.

The mesosigmoid and mesorectum are dissected from the right lateral rectum towards the root of the inferior mesenteric artery (IMA). The IMA is transected and ligated, so is the inferior mesenteric vein. Posterior space of the descending colon is dissected following opening the peritoneum beside the left rectum. The rectum in the pelvis is been mobilized from posterior rectal space, anterior rectal space to bilateral rectal space successively. The lower edge of the tumor is marked by a clamp. The linear stapler is placed in the pelvis to clamp the distal rectum below the tumor to see if the transection can be done more than 1cm from the lower edge of the tumor. If yes, the distal rectum will be transected by the traditional approach (that means the patient will be assigned to the traditional group). The proximal bowel is transected through a small midline incision. Then the coloanal anastomosis will be done intracorporeally. A surgical drain is placed in the pelvis and a terminal ileostomy is routinely performed. All incisions are closed.

If the distal rectal transection cannot be done more than 1cm from the lower edge of the tumor, the anterior obturator nerve gateway approach will be used (that means the patient will be assigned to the experimental group). The steps are as follows: The peritoneum covering the ureter and external iliac artery is opened more than 2 cm across the vas deferens (male) or round ligament (female). The Retzius space and vesicohypogastric fascia are exposed. The obturator vessels and obturator nerve are properly identified. Care should be taken to avoid any injury when using energy devices near the obturator nerve. The gateway is then opened through the TME (total mesorectal excision) compartment and the lateral compartment. If necessary, an "endoloop" can be placed through the gateway, and the bundled S2-4 nerves, ureter and bladder vessels are gently retracted toward the cranial direction to widen the gap. The linear stapler is placed in the gateway to vertically transect the distal rectum. The following procedures are the same with the traditional group as described above.

During the operation, the following variables will be recorded: the angle between the linear stapler and the rectum, distance from the lower edge to the resecting margin, whether the operation converted to transanal approach, operative time, bleeding volume, anastomotic height from anal verge and the length of the stapling line.

Postoperative management：

The following information will be recorded:

1）Vital signs (body temperature, pulse rate, respiration rate, blood pressure) are routinely monitored, gross volume of fluid input and output will be recorded every 24h, blood routine, the comprehensive metabolic panel and coagulation function tests will be performed every 3 days. 2）The time of catheter removal (days after operation), residual urine volume in the bladder will be measured by ultrasound examination. Whether there is a request to be re-catheterized or take oral medication to relive the dysuria. All patients will be asked to fulfil the IPSS (International prostate symptom score) questionnaire to assess urinary function. 3）The time of pelvic drain removal (days after operation). 4）Whether complicated with anastomotic leakage, ileus and long-lasting (more than 5 days) pulmonary or abdominal infection. 5）All information of the pathologic report. 6）Postoperative hospital stay (days) Postoperative chemoradiotherapy Radiotherapy program is the same with the neoadjuvant therapy. Chemotherapy will be advised for patients with stage II cancer accompanied with the following high-risk factors: histologically poorly differentiated with normal mismatched repair or stable microsatellite (MSS), pT4 (pathological stage T 4), vascular/nerve invasion, preoperative intestinal obstruction or perforation, ≤ 12 lymph nodes retrieved and R1 resection. The chemotherapy program is the same with neoadjuvant chemotherapy. If mismatch repair defect (dMMR) or high-level microsatellite instability (MSI-H) is confirmed by pathology, chemotherapy will not be advised. Patients with stage III cancer will routinely receive chemotherapy.

Follow-up

1) Information on general medical history and physical examination will be collected every 3 months for 3 years. 2) Blood tumor markers of CEA (carcinoembryonic antigen) and CA19-9 (carbohydrate antigen 19-9) will be tested every 3 months for 3 years. 3) Abdominal and pelvic ultrasound and chest X-ray examinations will be carried out every 3 months for 3 years. 4) Abdominal and pelvic MRI or contrast enhanced CT scan will be done every year for 3 years. 5) Colonoscopy will be performed within 1 year after surgery. If there is any abnormity, reexamination will be required within half a year. If no abnormality is found, once a year for 3 years. All new-found adenomas by the colonoscopy during follow-up are recommended to be resected. 6) Sexual function score is assessed by filling in the questionnaire (IIEF-5) both preoperatively and 1 year later since operation. 7) 3-year tumor-free survival (month): The time from operation to confirmation of tumor's local recurrence or distant metastasis. The end point of the patient lost to follow-up is the date of loss. 30 days is defined as one month. 8) 3-year overall survival (month): The time from operation to death. The end point of the patient lost to follow-up is the date of loss. 30 days is defined as one month. 9) Stoma closure time (months since operation). Anal function is assessed by Wexner scale 3 months and 12 months after stoma closure, respectively.

(As to possible risks and benefits of participating in this trial, see details in the informed consent document.) Study start date (actual) 2020-12-01 Study completion date (anticipated) 2025-12-01 (All outcomes of the last patient are recorded 3 years postoperatively, death or loss to follow-up of the last patient.) Statistics IBM SPSS (Statistical Package for the Social Sciences) Statistics 25 (IBM, Inc., Armonk, NY) will be used to perform statistical analyses. The t test and Mann-Whitney U test were used for quantitative data between groups. Qualitative data were compared by Chi-square test or Fisher's exact test and survival distributions were analyzed by log-rank test.

ELIGIBILITY:
Inclusion Criteria:

Pathologically diagnosed as rectal cancer with the lower margin of the tumor from the anal margin ≤5cm；CT, MRI or endoscopic ultrasonography: Single tumor, clinical T stage ≤3 or no invasion of the internal sphincter, maximum diameter ≤10cm, no distant metastasis；The patient or the patient-authorized representative completely understands the study protocol and voluntarily participates in this study, agrees to sign written informed consent.

Exclusion Criteria:

The patient had previous abdominal surgery that will significantly infect the laparoscopic procedures; Patients requiring emergency surgery owing to intestinal obstruction, perforation, or uncontrolled bleeding caused by tumor; Patients with poor anal function preoperatively (Wexner score ≥10); ASA (American Society of Anesthesiologists) grading ≥ IV; Pregnant patients; Patients concomitant with severe mental illness; The patient or the patient-authorized representative can't understand the contents and objectives of the study.

Withdraw criteria： ISR cannot be performed by intraoperative evaluation and is replaced by Miles surgery; Distant metastasis is confirmed intraoperatively or by postoperative pathological findings; Patients had other primary tumors requiring surgical/drug treatment during the study, or had other illnesses that prevent the patient from continuing to participate this study; Patients decide to withdraw from the study for any reason, or who are unable to complete the study because of any objective reasons.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
The degree of Angle | The degree of Angle will be measured on the resected specimen immediately after the surgery.
  The degree of angle between the linear stapler and the longitudinal axis of the rectum when transecting the distal rectum.
The degree of △Angle | The degree of △Angle will be measured on the resected specimen immediately after the surgery.
  The degree of angle between the simulated stapling line with the total mesorectal excision approach and the real stapling line with the transanterior obturator nerve gateway approach (this outcome is measured only in patients of the experimental group).
Length of distal resection margin | Length of distal resection margin will be measured by the operator immediately after the surgery and by the pathologist during the pathological test within a week after surgery, the final outcome will be the mean value of the two.
  The shortest distance between the distal border of the tumor and the edge of the distal resection.
Rate of conversion to transanal transection and anastomosis of the rectum. | The gross conversion rate will be calculated immediately after the last patient's surgery.
  The gross conversion rate (No. of cases undergoing conversion/total No. of cases enrolled *100%) will be calculated immediately after the last patient's surgery.
Rate of anastomotic leakage | For each case, whether complicated with anastomotic leakage will be supervised up to 6 months after surgery. The gross rate of anastomotic leakage will be calculated 6 months after the last patient's surgery.
  The gross anastomotic leakage rate (No. of cases diagnosed with anastomotic leakage/total No. of cases enrolled *100%) will be calculated 6 months after the last patient's surgery. Anastomotic leakage will be diagnosed if the patient has clinically apparent leakage signs (such as the emission of gas, pus, or feces from the pelvic drain, or peritonitis) or extravasation of endoluminally administered watersoluble contrast medium according to CT.

SECONDARY OUTCOMES:
Operative time | Operative time will be recorded immediately after the surgery.
  The time between the first incision and final closure of the operation.
Volume of blood loss | The gross volume of blood loss during the operation will be measured and recorded immediately after the surgery.
  The gross volume of blood loss during the operation.
Anastomotic height from anal verge | Anastomotic height will be measured and recorded by the operator using digital rectal exam immediately after the surgery.
  Distance between the coloanal anastomosis and the anal verge.
Length of stapling line | Length of stapling line will be measured directly on the resected specimen immediately after the surgery.
  The length of the lower stapling margin of the specimen.
Postoperative hospital stay | Postoperative hospital stay will be recorded on the day the patient is discharged from hospital.
  Days from operation to discharge from hospital.
Postoperative urinary retention in hospital | Whether there is urinary retention will be recorded before discharge from hospital or up to 30 days after surgery for each patient.
  Urinary retention is defined as requiring a second urinary catheterization or postvoid residual urine volume ≥ 50ml by ultrasound examination after first removal of the urinary catheter.
International prostate symptom score (IPSS) | Dysuria will be assessed by IPSS scale 1 month after surgery
  See IPSS scale in study protocol. Total score: 0-35 points, higher scores mean worse outcome.
Wexner score | Anal function evaluated by Wexner score will be assessed 3 and 12 months after stoma closure
  See Wexner score in study protocol. Total score: 0-20 points, higher scores mean worse outcome.
International Index of Erectile Function (IIEF-5) score | Sexual function will be assessed by IIEF-5 scale 1 week before surgery and 12 months after surgery
  See IIEF-5 scale in study protocol. Total score: 5-25 points, higher scores mean better outcome.
3-year overall survival | Survival information after 3 years from operation or till death/loss of follow-up within 3 years from operation will be collected for each patient.
  The percentage of people who are alive after 3 years from operation.
3-year disease-free survival | Survival without cancer relapse or metastasis after 3 years from operation or till cancer relapse/metastasis/death/loss of follow-up within 3 years from operation will be recorded for each patient.
  The percentage of patients who are alive without cancer relapse or metastasis after 3 years from operation.

CONTACTS AND LOCATIONS:
Overall Officials: Jianqiang Tang, MD, Study Chair — Peking University First Hospital
Locations (4):
- China (4):
  - The Second Affiliated Hospital of Baotou Medical University, Baotou, Inner Mongolia
  - Dalian University Affiliated Xinhua Hospital, Dalian, Liaoning
  - Shengli Oilfield Hospital, Dongying, Shandong
  - The Third People's Hospital of Datong, Datong, Shanxi

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Background] Scala D, Niglio A, Pace U, Ruffolo F, Rega D, Delrio P. Laparoscopic intersphincteric resection: indications and results. Updates Surg. 2016 Mar;68(1):85-91. doi: 10.1007/s13304-016-0351-6. Epub 2016 Mar 29. PMID 27022927
- [Background] Chi P, Huang SH, Lin HM, Lu XR, Huang Y, Jiang WZ, Xu ZB, Chen ZF, Sun YW, Ye DX. Laparoscopic transabdominal approach partial intersphincteric resection for low rectal cancer: surgical feasibility and intermediate-term outcome. Ann Surg Oncol. 2015 Mar;22(3):944-51. doi: 10.1245/s10434-014-4085-8. Epub 2014 Sep 23. PMID 25245128
- [Background] Fujimoto Y, Akiyoshi T, Kuroyanagi H, Konishi T, Ueno M, Oya M, Yamaguchi T. Safety and feasibility of laparoscopic intersphincteric resection for very low rectal cancer. J Gastrointest Surg. 2010 Apr;14(4):645-50. doi: 10.1007/s11605-009-1150-x. Epub 2010 Jan 22. PMID 20094813
- [Background] Braun J, Treutner KH, Winkeltau G, Heidenreich U, Lerch MM, Schumpelick V. Results of intersphincteric resection of the rectum with direct coloanal anastomosis for rectal carcinoma. Am J Surg. 1992 Apr;163(4):407-12. doi: 10.1016/0002-9610(92)90042-p. PMID 1532699
- [Background] Pai VD, Sugoor P, Patil PS, Ostwal V, Engineer R, Arya S, Desouza A, Saklani AP. Laparoscopic Versus Open Approach for Intersphincteric Resection-Results from a Tertiary Cancer Center in India. Indian J Surg Oncol. 2017 Dec;8(4):474-478. doi: 10.1007/s13193-017-0672-z. Epub 2017 Jun 21. PMID 29203976
- [Background] Mahalingam S, Seshadri RA, Veeraiah S. Long-Term Functional and Oncological Outcomes Following Intersphincteric Resection for Low Rectal Cancers. Indian J Surg Oncol. 2017 Dec;8(4):457-461. doi: 10.1007/s13193-016-0571-8. Epub 2016 Oct 28. PMID 29203973
- [Background] Denost Q, Rullier E. Intersphincteric Resection Pushing the Envelope for Sphincter Preservation. Clin Colon Rectal Surg. 2017 Nov;30(5):368-376. doi: 10.1055/s-0037-1606114. Epub 2017 Nov 27. PMID 29184472
- [Background] Park SY, Choi GS, Park JS, Kim HJ, Ryuk JP. Short-term clinical outcome of robot-assisted intersphincteric resection for low rectal cancer: a retrospective comparison with conventional laparoscopy. Surg Endosc. 2013 Jan;27(1):48-55. doi: 10.1007/s00464-012-2405-2. Epub 2012 Jun 30. PMID 22752275
- [Background] Bi L, Deng X, Meng X, Yang X, Wei M, Wu Q, Ren M, Wang Z. Ligating the rectum with cable tie facilitates rectum transection in laparoscopic anterior resection of rectal cancer. Langenbecks Arch Surg. 2020 Mar;405(2):233-239. doi: 10.1007/s00423-020-01863-6. Epub 2020 Apr 8. PMID 32266529
- [Background] Hotta T, Takifuji K, Yokoyama S, Matsuda K, Oku Y, Hashimoto T, Yamamoto N, Yamaue H. Rectal transection by the Nelaton catheter pulling method during a laparoscopic low anterior resection. Dis Colon Rectum. 2011 Apr;54(4):495-500. doi: 10.1007/DCR.0b013e318207026f. PMID 21383572
- [Background] Park SJ, Choi SI, Lee SH, Lee KY. Endo-satinsky clamp for rectal transection during laparoscopic total mesorectal excision. Dis Colon Rectum. 2010 Mar;53(3):355-9. doi: 10.1007/DCR.0b013e3181c388e9. PMID 20173486
- [Background] Brannigan AE, De Buck S, Suetens P, Penninckx F, D'Hoore A. Intracorporeal rectal stapling following laparoscopic total mesorectal excision: overcoming a challenge. Surg Endosc. 2006 Jun;20(6):952-5. doi: 10.1007/s00464-005-0536-4. Epub 2006 May 12. PMID 16738989

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-09-07): https://cdn.clinicaltrials.gov/large-docs/13/NCT05067413/Prot_SAP_ICF_000.pdf